CLINICAL TRIAL: NCT06515873
Title: Evaluating the Acceptability of Virtual Reality Headsets During Surgery Under Spinal Anesthesia in Elderly Patients. Seniors' Intraoperative Management Under Locoregional Anesthesia Integrating Virtual Reality (SILVR)
Brief Title: Seniors' Intraoperative Management Under Locoregional Anesthesia Integrating Virtual Reality
Acronym: SILVR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Pascal Laferrière-Langlois, MD, MSc, FRQS, Assistant Professor, Principal Investigator, Anesthesiologist, Ciusss de L'Est de l'Île de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-3770
Record Dates: First submitted 2024-07-11; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Virtual Reality; Spinal Anesthesia
Keywords: Elderly patient; Acceptability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a group of 55 patients (Experimental)
  Interventions: Device: Virtual Reality Headset

INTERVENTIONS:
Device: Virtual Reality Headset — The virtual reality headset, which will display one of the 3 available scenarios, will be placed on the patient head during a surgery under spinal anesthesia.

SUMMARY:
This study aims to evaluate the acceptability of intraoperative virtual reality in elderly patients under spinal anesthesia.

DETAILED DESCRIPTION:
For the past decade, virtual reality (VR) has been expanding across various medical applications fields. Regarding surgery and anesthesia, VR was used during different procedures such as orthopedics surgery of the upper extremities under regional anesthesia blocks, hip and knee arthroplasties, dental care and induction of anesthesia, especially in pediatrics. Using VR during surgery can reduce pain, anxiety, quantity of sedation used and time in the PACU.

Unfortunately, the adherence to VR specifically among adults aged 65 and over is not thoroughly defined in the scientific literature and should be investigated in order to determine the spectrum of use of this tool. However, VR has been used as an anxiolytic and analgesic in elderly patients during rehabilitation exercises, such as physiotherapy treatment after surgery or vestibular rehabilitation after experiencing dizziness.

The main objective of this study is to determine if a virtual reality headset can be tolerated during surgery under spinal anesthesia in patients aged 65 years and older. 55 patients over 65 years old having an elective surgery will be recruited.

The total time for which the patient will wear the virtual reality headset during the surgery will be measured and a semi-structured post-operative questionnaire will assess the overall patient satisfaction.

Simultaneously, the influence of the type of scenario chosen on the patient's tolerance to the VR headset will be established (secondary objective details listed below)

Study Center: Maisonneuve-Rosemont Hospital, Integrated University Health and Social Services Centre (CIUSSS) de l'Est de l'Ile de Montreal (CEMTL), University of Montreal, Montreal, Quebec, Canada

ELIGIBILITY:
Inclusion Criteria:

* Fully consented patients over 65 years old
* Undergoing elective surgery that requires spinal anesthesia.

Exclusion Criteria:

* Hearing or visual impairment
* History of epilepsy, seizure, or severe dizziness
* Severe mental impairment
* Recent eye or facial surgery or wounds
* Inability to use their hands

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Patient's tolerance to headset | Intraoperative (from T0 = the patient puts on the headset until Tend = 30 minutes after T0)
  The primary endpoint is the patient's tolerance to virtual reality defined by the headset to be worn for more than or equal to 30 minutes by the participant

SECONDARY OUTCOMES:
Anxiety before the surgery | preoperative (from T0 = the patient arrives at the hospital the morning of the surgery until Tend = the patient enters the operating room, about 2 hours)
  Level of anxiety before the surgery evaluated by the Amsterdam Preoperative Anxiety and Information Scale (a scale from 1 - not at all to 5 - extremely, 6 questions).
Total of time before the patient's first request to interrupt the experiment | intraoperative (from T0 = the patient puts on the headset at the beginning of the surgery until Tend = the patient first asks to interrupt the experiment during the surgery, about 45 minutes - depending on the person and the surgery)
  The total time in minutes, both in absolute and relative to the duration of the surgery, from the start of the initially chosen scenario to the first request to interrupt the experiment.
Total of time during which the patient wears the VR headset during surgery. | intraoperative (from T0 = the patient puts on the headset and starts the initially chosen scenario until Tend = the patient takes off the headset, about 45 minutes - depending on the person and the surgery)
  The total time in minutes, both in absolute and relative to the duration of the surgery, from the start of the initially chosen scenario to the headset removal
Time spent on each scenario and the order in which they were presented | intraoperative (from T0 = the patient starts the first scenario until Tend = he asks to change the scenario) - for each scenario, about 45 minutes - depending on the person and the surgery
  Compare the total duration in minutes the patient wore the headset depending on the type of scenario chosen, and the order in which they were presented
Incidence of adverse effects | intraoperative (from T0 = the patient puts on the headset until Tend = the patient takes off the headset, about 45 minutes - depending on the surgery)
  The incidence of adverse effects such as cybersickness, as reported by the patient
Patient's satisfaction | postoperative (from T0 = the surgery ends until Tend = the semi-structured questionnaire is over, about 2 hours)
  The satisfaction, ease to use the VR and main complaints of the participant, assessed through interviews using semi-standardized questions (17 open questions during a discussion, transcribe verbatim, to make a qualitative analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Laferrière-Langlois, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Maisonneuve-Rosemont Hospital - CIUSSS de l'Est de l'Île de Montréal, Montreal East, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boutin J, Kamoonpuri J, Faieghi R, Chung J, de Ribaupierre S, Eagleson R. Smart haptic gloves for virtual reality surgery simulation: a pilot study on external ventricular drain training. Front Robot AI. 2024 Jan 10;10:1273631. doi: 10.3389/frobt.2023.1273631. eCollection 2023. PMID 38269073
- [Background] Boyce L, Jordan C, Egan T, Sivaprakasam R. Can virtual reality enhance the patient experience during awake invasive procedures? A systematic review of randomized controlled trials. Pain. 2024 Apr 1;165(4):741-752. doi: 10.1097/j.pain.0000000000003086. Epub 2023 Oct 23. PMID 37870233
- [Background] Eijlers R, Utens EMWJ, Staals LM, de Nijs PFA, Berghmans JM, Wijnen RMH, Hillegers MHJ, Dierckx B, Legerstee JS. Systematic Review and Meta-analysis of Virtual Reality in Pediatrics: Effects on Pain and Anxiety. Anesth Analg. 2019 Nov;129(5):1344-1353. doi: 10.1213/ANE.0000000000004165. PMID 31136330
- [Background] Fuchs L, Kluska A, Novak D, Kosashvili Y. The influence of early virtual reality intervention on pain, anxiety, and function following primary total knee arthroplasty. Complement Ther Clin Pract. 2022 Nov;49:101687. doi: 10.1016/j.ctcp.2022.101687. Epub 2022 Nov 5. PMID 36347152
- [Background] Hitching R, Hoffman HG, Garcia-Palacios A, Adamson MM, Madrigal E, Alhalabi W, Alhudali A, Sampaio M, Peterson B, Fontenot MR, Mason KP. The Emerging Role of Virtual Reality as an Adjunct to Procedural Sedation and Anesthesia: A Narrative Review. J Clin Med. 2023 Jan 20;12(3):843. doi: 10.3390/jcm12030843. PMID 36769490
- [Background] Huang MY, Scharf S, Chan PY. Effects of immersive virtual reality therapy on intravenous patient-controlled sedation during orthopaedic surgery under regional anesthesia: A randomized controlled trial. PLoS One. 2020 Feb 24;15(2):e0229320. doi: 10.1371/journal.pone.0229320. eCollection 2020. PMID 32092098
- [Background] Kanyilmaz T, Topuz O, Ardic FN, Alkan H, Oztekin SNS, Topuz B, Ardic F. Effectiveness of conventional versus virtual reality-based vestibular rehabilitation exercises in elderly patients with dizziness: a randomized controlled study with 6-month follow-up. Braz J Otorhinolaryngol. 2022 Nov-Dec;88 Suppl 3(Suppl 3):S41-S49. doi: 10.1016/j.bjorl.2021.08.010. Epub 2021 Oct 26. PMID 34799265
- [Background] Kuhn AW, Yu JK, Gerull KM, Silverman RM, Aleem AW. Virtual Reality and Surgical Simulation Training for Orthopaedic Surgery Residents: A Qualitative Assessment of Trainee Perspectives. JB JS Open Access. 2024 Mar 20;9(1):e23.00142. doi: 10.2106/JBJS.OA.23.00142. eCollection 2024 Jan-Mar. PMID 38511201
- [Background] Roxburgh T, Li A, Guenancia C, Pernollet P, Bouleti C, Alos B, Gras M, Kerforne T, Frasca D, Le Gal F, Christiaens L, Degand B, Garcia R. Virtual Reality for Sedation During Atrial Fibrillation Ablation in Clinical Practice: Observational Study. J Med Internet Res. 2021 May 27;23(5):e26349. doi: 10.2196/26349. PMID 34042589
- [Background] Ryu S, Kitagawa T, Goto K, Okamoto A, Marukuchi R, Hara K, Ito R, Nakabayashi Y. Intraoperative Holographic Guidance Using Virtual Reality and Mixed Reality Technology During Laparoscopic Colorectal Cancer Surgery. Anticancer Res. 2022 Oct;42(10):4849-4856. doi: 10.21873/anticanres.15990. PMID 36192000
- [Background] Wang Y, Guo L, Xiong X. Effects of Virtual Reality-Based Distraction of Pain, Fear, and Anxiety During Needle-Related Procedures in Children and Adolescents. Front Psychol. 2022 Apr 19;13:842847. doi: 10.3389/fpsyg.2022.842847. eCollection 2022. PMID 35519646
- [Background] Yi WS, Rouhi AD, Duffy CC, Ghanem YK, Williams NN, Dumon KR. A Systematic Review of Immersive Virtual Reality for Nontechnical Skills Training in Surgery. J Surg Educ. 2024 Jan;81(1):25-36. doi: 10.1016/j.jsurg.2023.11.012. Epub 2023 Nov 30. PMID 38036388